CLINICAL TRIAL: NCT00733928
Title: Randomised Prospective Comparison of P.F.C All-polyethylene Versus Metal-backed Tibial Component. A Clinical, Radiological and Roentgen Stereophotogrammetric Analysis (RSA) Study.
Brief Title: The Press Fit Condylar (P.F.C.) Sigma Metal-backed Versus All-poly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT 99/26
Record Dates: First submitted 2008-08-11; First posted 2008-08-13 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis
Keywords: Arthroplasty,; Replacement,; Knee,; P.F.C.; Sigma; all-polyethylene
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 - All Polyethylene Tibia (Other): Total knee replacement with an all polyethylene tibial tray
  Interventions: Device: PFC Sigma knee with all-poly tibial component
- 2 - Poly & Metal Tibia (Active Comparator): Total knee replacement with a metal-backed tibial component
  Interventions: Device: PFC Sigma knee with metal backed tibia

INTERVENTIONS:
Device: PFC Sigma knee with all-poly tibial component — Orthopaedic implant for total knee replacement with an all-polyethylene tibial component
  Arms: 1 - All Polyethylene Tibia
Device: PFC Sigma knee with metal backed tibia — Orthopaedic implant for total knee replacement with a metal-backed tibial component
  Arms: 2 - Poly & Metal Tibia

SUMMARY:
The primary objective of this investigation was to evaluate & compare the performance of the P.F.C. Sigma Knee Cruciate-retaining all-polyethylene and metal-backed tibia components using RSA.

The secondary objectives of this investigation are to evaluate the clinical and patient outcomes and survivorship associated with the P.F.C. Sigma Knee Cruciate-retaining all-polyethylene and metal-backed tibia components.

DETAILED DESCRIPTION:
Using RSA, is it possible to evaluate the performance of both the all polyethylene and metal backed tibia components to determine whether there are differences in migration, if present, across the tibial components.

The original protocol intended to perform clinical assessment using the Nottingham Knee Score and the Knee Society Clinical rating system pre-and post-operatively, at six months, 1 year, and annually thereafter. Per Protocol Amendment 01 (effective June 18, 1999) clinical data would also be collected via the SF-12 questionnaire. Radiological evaluation would also use the Knee Society scoring system at the same time points. However, data collected included only the SF-12 and Oxford Knee Scores, comparing change from baseline at 6, 12, and 24 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects requiring a primary knee replacement.
* Subjects aged 65 years or more.
* Subjects who are able to give voluntary, written informed consent to participate in this clinical investigation and from whom consent has been obtained.
* Subjects with a primary diagnosis of osteoarthritis or rheumatoid arthritis.

Exclusion Criteria:

* Subjects who have had a previous surgery of the operative knee except menisectomy and arthroscopy.
* Subjects who have had a renal transplant.
* Subjects with a metabolic bone disorder.
* Subjects who, in the opinion of the Clinical Investigator, have an existing condition, e.g. Paget's disease etc. that would compromise their participation and follow-up in this clinical investigation.
* Subjects whose contralateral knee is already included in this study.
* Subjects who have a history of active joint sepsis.
* Subjects who have a recent history of high dose systemic corticosteroids.
* Subjects with psycho-social disorders or physical disabilities that would limit rehabilitation.
* Subjects requiring a bone graft.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 67 (Actual)
Dates: Start 1999-10-01 (Actual); Primary Completion 2005-05-01 (Actual); Study Completion 2015-03-01 (Actual)

PRIMARY OUTCOMES:
Using RSA it is possible to evaluate the performance of both the all-polyethylene and metal-backed tibia components to determine whether there are differences in migration between the two components | 2 years

SECONDARY OUTCOMES:
Comparative evaluation of any post-operative variation between subjects receiving all-polyethylene and metal-backed tibia components in change from baseline at each post operative time points in terms of SF 12 and OKS | 6 months, 1 year and 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics, Freeman Hospital, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Result] Muller SD, Deehan DJ, Holland JP, Outterside SE, Kirk LM, Gregg PJ, McCaskie AW. Should we reconsider all-polyethylene tibial implants in total knee replacement? J Bone Joint Surg Br. 2006 Dec;88(12):1596-602. doi: 10.1302/0301-620X.88B12.17695. PMID 17159170